CLINICAL TRIAL: NCT06046924
Title: Dietary Acid Reduction and Progression of Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-INTMED-95987
Record Dates: First submitted 2023-08-16; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Chronic Kidney Diseases; Cardiovascular Diseases; Hypertension
Keywords: albuminuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Hypertension; Albuminuria | interventions — Fruit; Vegetables; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fruits and vegetables (F+V) (Experimental): 51 participants with hypertension, normal estimated glomerular filtration rate (eGFR) (>90 ml/min/m2) and macroalbuminuria (albumin [mg] to creatinine [g] ratio > 200 mg/g) will receive a prescribed amount of base-producing fruits and vegetables (F+V) designed to reduce their dietary acid intake by half. Depending on the particular foods used, this amounts to 2-4 cups daily of fruits and vegetables given in weekly allotments. They will otherwise receive standard care for their medical concerns including angiotensin converting enzyme inhibitor therapy for albuminuria and followed annually for 5 years.
  Interventions: Other: Fruits and vegetables (F+V)
- NaHCO3 (HCO3) (Experimental): 51 participants with hypertension, normal estimated glomerular filtration rate (eGFR) (>90 ml/min/m2) and macroalbuminuria (albumin [mg] to creatinine [g] ratio > 200 mg/g) will receive 0.4 mEq/kg/bw oral tablet dose of sodium bicarbonate (NaHCO3) designed to match the alkali intake of F+V. They will otherwise receive standard care for their medical concerns including angiotensin converting enzyme inhibitor therapy for albuminuria and followed annually for 5 years.
  Interventions: Drug: NaHCO3 Tablets
- Usual Care (UC) (Active Comparator): 51 participants with hypertension, normal estimated glomerular filtration rate (eGFR) (>90 ml/min/m2) and macroalbuminuria (albumin [mg] to creatinine [g] ratio > 200 mg/g) will receive no additional alkali (neither F+V or NaHCO3) and will receive standard care for their medical concerns, including angiotensin converting enzyme inhibitor therapy for albuminuria and followed annually for 5 years.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Fruits and vegetables (F+V) — Participants will receive a prescribed amount of F+V designed to reduce their dietary acid intake by half. This typically amounts to 2-4 cups/day for each participant randomized to this group, depending on the type of F+Vs used, provided in weekly allotments. Participants will receive standard care for their medical concerns.
  Arms: Fruits and vegetables (F+V)
Drug: NaHCO3 Tablets — Participants will receive 0.4 mEq/kg bw NaHCO3 /day, an amount designed to match the alkali provided by the added F+V. This will be provided as 650 mg NaHCO3 tablets for an average of 4-5 tablets/day in 2 divided doses for each participant randomized to this group. Participants will receive standard care for their medical concerns.
  Other Names: Baking soda
  Arms: NaHCO3 (HCO3)
Other: Usual Care — Participants will receive standard care for their medical concerns and no additional alkali (F+V or NaHCO3).
  Arms: Usual Care (UC)

SUMMARY:
Upon completion, this project will determine if dietary acid reduction done with either fruits and vegetables (F+V) or the medication sodium bicarbonate (NaHCO3) in study participants with high blood pressure (hypertension) and initially normal kidney function but with signs of kidney injury 1) slows progression of chronic kidney disease (CKD); 2) improves indices of cardiovascular risk; and 3) better preserves acid-base status. These studies are designed to determine if the simple and comparatively inexpensive intervention of dietary acid reduction can prevent or reduce adverse outcomes in individuals with early-stage CKD.

DETAILED DESCRIPTION:
The long-term objective of this study is to determine if the simple and comparatively inexpensive intervention of dietary acid reduction can prevent or reduce adverse outcomes in individuals with hypertension and early-stage chronic kidney disease (CKD). The specific aims of this study are to determine if dietary acid reduction done with either base-producing fruits and vegetables (F+V) in amounts calculated to reduce participant dietary acid content by half or with sodium bicarbonate (NaHCO3, 0.4 milliequivalents (mEq)/kg body weight (bw), an amount designed to match the alkali content of the prescribed F+V) in participants with initially normal kidney function but with signs of kidney injury 1) slows progression of CKD; 2) improves indices of cardiovascular risk; and 3) better preserves acid-base status. The incidence and prevalence of CKD is increasing along with increased incidence and prevalence of its adverse outcomes, including heart attack and stroke, the latter for which patients with CKD are at increased risk. Most modern diets produce acid when metabolized in the body and some studies suggest that the small amount of acid produced causes progressive and long-term injury to blood vessels in kidneys, heart, and brain, thereby increasing risk for kidney disease and its progression, heart attack and stroke. This study will recruit participants with hypertension and macroalbuminuria (urine albumin [mg]-to-creatinine [g] ratio > 200 mg/g) but with normal estimated glomerular filtration rate (eGFR) greater than or equal to 90 ml/min/1.73 m2) to be randomized to receive dietary acid reduction done with F+V or oral NaHCO3 or to no dietary acid reduction (Usual Care). At study entry and yearly for 5 years, all participants will have 10 milliliters (ml) of blood drawn from an antecubital vein for measurement of pH, partial pressure of carbon dioxide (PCO2), total CO2 (TCO2), creatinine, cystatin-C, low-density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholesterol, Lp(a) cholesterol, sodium, potassium, chloride, and citrate. They will also have 20 ml of urine collected for measurement of creatinine, pH, TCO2, ammonium, titratable acidity, albumin, N-acetyl-D-glucosaminidase, angiotensinogen, isoprostane 8-isoprostaglandin F2 alpha (8-iso), and citrate. Body acid will be measured in participants at baseline and at 5 years during an 8-hour protocol conducted in a Texas Tech University Health Sciences Center (TTUHSC) clinic. They will be told to fast after midnight and report to the TTUHSC clinic the following morning at which time they will be given a single oral dose of sodium bicarbonate (NaHCO3, 0.5 mEq/kg) and have 1 ml of blood drawn from a needle maintained in an arm vein for protocol duration for TCO2 before and at 2, 4, and 6 hours after the dose of NaHCO3 was given and urine collected over 8 hours for TCO2, pH, ammonium, and titratable acidity. The change in blood TCO2 in response to the amount of bicarbonate retained the body (dose minus urine bicarbonate excretion) will be used to calculate participant body acid. The course of serum and urine parameters over the 5 years of follow up in those randomized to F+V or NaHCO3 compared to Usual Care will help determine the effect of dietary acid reduction on CKD progression (change in eGFR and in urine indices of kidney injury), indices of cardiovascular disease risk (change in LDL, HDL, and Lp(a) cholesterol, and change in 8-iso), and on participant acid-base status (serum acid-base parameters (pH, PCO2, bicarbonate concentration [HCO3], TCO2, urine citrate excretion, and body acid measurement). These studies will also determine differences in these outcomes with dietary acid reduction done with F+V or NaHCO3.

The investigators hypothesize that dietary acid reduction will 1) reduce kidney injury indicated by lower urine indices of kidney injury and slow kidney function decline indicated by slower eGFR decline rate; 2) improve indices of cardiovascular risk indicated by lower LDL, higher HDL, lower Lp(a) cholesterol, and lower 8-iso; and 3) improve acid-base status indicated by higher serum TCO2, higher urine citrate excretion, and lower body acid. The investigators additionally hypothesize that F+V will have greater benefits on indicators of parameters of cardiovascular risk than NaHCO3. Excretion of urine acid-base parameters will help determine effects of dietary acid reduction on urine acid excretion. Blood pH and PCO2 will be measured using a blood gas analysis system and blood and urine concentrations of albumin and creatinine will be measured with standard techniques. Blood and urine TCO2 will be measured as done previously using fluorimetry techniques in the PI's laboratory. Urine ammonium, titratable acidity, N-Acetyl-beta-D-glucosaminidase, angiotensinogen, isoprostane 8-isoprostaglandin F2 alpha and citrate will be measured as done previously in the laboratory of the Co-PI.

ELIGIBILITY:
Inclusion Criteria:

* Non-malignant high blood pressure or hypertension
* 18-70 years old
* Urine albumin-to-creatine ratio > 200 mg/g creatinine
* Estimated glomerular filtration rate (eGFR) greater than or equal to 90 ml/min/1.73 m2
* Serum total CO2 (TCO2) > 22 mmol/l
* Greater than or equal to 2 primary care visits in the preceding year
* Able to provide informed consent

Exclusion Criteria:

* Malignant hypertension or history thereof
* Primary kidney disease or findings consistent thereof such as > 3 red blood cells per high powered field of urine or urine cellular casts
* History of diabetes or fasting glucose greater than or equal to 110 mg/dl
* History of hematologic disorders, malignancies, chronic infections, current pregnancy, history or clinical evidence of cardiovascular disease
* Peripheral edema or diagnosis associated with edema such as heart/liver failure or nephrotic syndrome
* Unable to provide consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 1996-06-24 (Actual); Primary Completion 2006-11-15 (Actual); Study Completion 2011-12-15 (Actual)

PRIMARY OUTCOMES:
Difference in estimated glomerular filtration rate (eGFR) at 5 years follow up | eGFR will be measured at baseline and yearly for 5 years.
  eGFR (ml/min/1.73 m2) will be calculated using measured serum creatinine and cystatin-C concentrations, age, sex, and whether or not of African American ethnicity using a standard accepted formula.
  eGFR will be compared among the three groups at 5 years follow up to assess chronic kidney disease (CKD) progression. Higher eGFR is indicative of better-preserved kidney function. The investigators hypothesize that dietary acid reduction will lead to better preserved (higher) eGFR at 5 years.
Difference in the rate of eGFR change during 5 years follow up | eGFR will be measured at baseline and yearly for 5 years.
  The rate of eGFR change (ml/min/1.73 m2/year) will assess CKD progression and will be calculated by dividing the net change in eGFR over 5 years (5-year value minus baseline value) and dividing by 5 years. The investigators hypothesize that dietary acid reduction will lead to a slower rate of eGFR change, indicative of less CKD progression.
Difference in the net eGFR change during 5 years follow up | eGFR will be measured at baseline and yearly for 5 years.
  The net eGFR change (ml/min/1.73 m2) will assess CKD progression and will be calculated by subtracting the 5-year value from the baseline value. The investigators hypothesize that dietary acid reduction will lead to a smaller net eGFR change, indicative of less CKD progression.
Difference in change in urine albumin excretion during 5 years follow up | ACR will be measured at baseline and yearly for 5 years.
  CKD progression will be assessed by change in the albumin (mg)-to-creatinine (g) ratio (ACR) in a "spot" urine. An increased ACR is indicative of kidney injury and risk for subsequent decrease of kidney function with time. A decrease in ACR is indicative of reduced kidney injury and a lower risk for decreased kidney function with time. The investigators hypothesize that dietary acid reduction will lead to a lower ACR.
  • ACR will be compared among the three groups as follows:
  * 5 year value
  * Net change (5 year value minus baseline value) at five years
Difference in change in urine N-acetyl-D -glucosaminidase (NAG) excretion during 5 years follow up | NAG/creatinine will be measured at baseline and yearly for 5 years.
  CKD progression will be assessed by change in the NAG (Units)-to-creatinine (g) ratio in a "spot" urine. An increased NAG/creatinine ratio is indicative of increased kidney injury. The investigators hypothesize that dietary acid reduction will lead to a lower NAG/creatinine.
  • NAG/creatinine will be compared among the three groups as follows:
  * 5 year value
  * Net change (5 year value minus baseline value) at five years
Difference in change in urine angiotensinogen (ATG) excretion during 5 years follow up | ATG/creatinine will be measured at baseline and yearly for 5 years.
  CKD progression will be assessed by change in the ATG (ug)-to-creatinine (g) ratio in a "spot" urine. An increased ATG/creatinine ratio is an indirect measure of kidney levels of angiotensin II and is indicative of increased kidney injury. The investigators hypothesize that dietary acid reduction will lead to a lower ATG/creatinine ratio.
  • ATG/creatinine will be compared among the three groups as follows:
  * 5 year value
  * Net change (5 year value minus baseline value) at five years

SECONDARY OUTCOMES:
Difference in change in serum LDL cholesterol level during 5 years follow up | Serum LDL cholesterol will be measured at baseline and yearly for 5 years.
  Higher serum LDL cholesterol levels (mg/dl) are an indicator of increased cardiovascular disease risk. The investigators hypothesize that dietary acid reduction done with fruits and vegetables leads to lower LDL cholesterol than that done with either sodium bicarbonate or Usual Care.
  Comparisons among the three groups will be done as follows:
  1. level at 5 years
  2. Net change at 5 years
Difference in change in serum HDL cholesterol level during 5 years follow up | Serum HDL cholesterol will be measured at baseline and yearly for 5 years.
  Higher serum HDL cholesterol levels (mg/dl) are an indicator of decreased cardiovascular disease risk. The investigators hypothesize that dietary acid reduction done with fruits and vegetables leads to higher LDL cholesterol than that done with either sodium bicarbonate or Usual Care.
  Comparisons among the three groups will be done as follows:
  1. level at 5 years
  2. Net change at 5 years
Difference in change in serum Lp(a) cholesterol level during 5 years follow up | Serum Lp(a) cholesterol will be measured at baseline and yearly for 5 years.
  Higher serum Lp(a) cholesterol levels (mg/dl) are an indicator of increased cardiovascular disease risk. The investigators hypothesize that dietary acid reduction done with fruits and vegetables leads to lower Lp(a) cholesterol than that done with either sodium bicarbonate or Usual Care.
  Comparisons among the three groups will be done as follows:
  1. level at 5 years
  2. Net change at 5 years
Difference in change in urine Isoprostane 8-isoprostaglandin F2α excretion during 5 years follow up | Urine Isoprostane 8-isoprostaglandin F2α to creatinine ratio will be measured at baseline and yearly for 5 years.
  Higher urine excretion of Isoprostane 8-isoprostaglandin F2α (8-iso) is an indicator of increased oxidative stress which contributes to increased cardiovascular disease risk. It will be measured as 8-iso (ug)-to-creatinine (g) ratio in a "spot" urine. The investigators hypothesize that dietary acid reduction leads to a lower 8-iso/creatinine ratio.
  Comparisons among the three groups will be done as follows:
  1. level at 5 years
  2. Net change at 5 years
Difference in change in serum pH during 5 years follow up | Serum pH will be measured at baseline and yearly for 5 years.
  Serum pH (pH is expressed numerically without units) will be measured with standard blood gas machine techniques. The investigators hypothesize that dietary acid reduction will lead to higher values for serum pH.
  Comparisons among the three groups will be as follows:
  * Levels at five years
  * Net change at five years
Difference in change in serum partial pressure of carbon dioxide gas (PCO2) during 5 years follow up | Serum PCO2 will be measured at baseline and yearly for 5 years.
  Serum PCO2 [millimeter (mm) mercury (Hg)], will be measured with standard blood gas machine techniques. The investigators hypothesize that dietary acid reduction will lead to higher values for serum PCO2.
  Comparisons among the three groups will be as follows:
  * Levels at five years
  * Net change at five years
Difference in change in serum bicarbonate concentration (HCO3-]) during 5 years follow up | Serum [HCO3-] will be measured at baseline and yearly for 5 years.
  Serum [HCO3-] (mEq/l) will be calculated from measured values of serum pH and serum partial pressure of carbon dioxide gas (PCO2) with a conventional formula commonly used by clinical laboratories. The investigators hypothesize that dietary acid reduction will lead to higher values for serum [HCO3-].
  Comparisons among the three groups will be as follows:
  * Levels at five years
  * Net change at five years
Difference in change in serum total CO2 (TCO2) during 5 years follow up | Serum TCO2 will be measured at baseline and at 5 years.
  TCO2 [millimolar (mM)] will be measured by the PI as in previous studies using ultrafluorimetry. This technique uses an enzymatic assay in which TCO2 reacts with phosphoenolpyruvate to form oxaloacetate, which is reduced to malate coupled with oxidation of nicotinamide adenine dinucleotide bound to hydrogen ion (NADH) to nicotinamide adenine dinucleotide without hydrogen ion (NAD+). NADH fluoresces but NAD+ does not, allowing for quantitation of TCO2 as reduced fluorescence. This technique is more reproducible than the conventional one of measuring CO2 gas released upon addition of a strong acid.
  Measuring changes in serum TCO2 will help assess the effect(s) of dietary acid reduction among the three groups. The investigators hypothesize that dietary acid reduction will lead to higher values for serum TCO2.
  Comparisons among the three groups will be as follows:
  * Levels at five years
  * Net change at five years
Difference in change in serum citrate concentration during 5 years follow up | Serum citrate will be measured at baseline and yearly for 5 years.
  Urine citrate excretion (millimoles [mmoles]/8 hours) will be measured to assess acid base status. Higher urine citrate excretion is indicative of lower body acid. The investigators hypothesize that dietary acid reduction will lead to greater urine citrate excretion.
  Comparisons among the three groups will be as follows:
  * Level at five years
  * Net change at five years
Difference in change in urine citrate excretion during 5 years follow up | Urine citrate excretion will be measured at baseline and yearly for 5 years.
  Urine citrate excretion (millimoles [mmoles]/8 hours) will be measured to assess acid base status. Higher urine citrate excretion is indicative of lower body acid. The investigators hypothesize that dietary acid reduction will lead to greater urine citrate excretion.
  Comparisons among the three groups will be as follows:
  * Level at five years
  * Net change at five years
Difference in change in body acid retention during 5 years follow up | Acid retention will be measured at baseline and at 5 years.
  This technique for body acid assessment was originated by the PI.
  Participants will have venous blood drawn for TCO2, receive oral NaHCO3 (0.5 mEq/kg lean bw), and have venous blood drawn for TCO2 at 2, 4, and 6 hours (4 total blood samples) after the NaHCO3 dose. All urine excreted over 8 hours will be collected to determine the amount of urine HCO3 excreted estimated by measuring urine TCO2. Body acid retention will be calculated as the difference between expected (retained HCO3-/HCO3- space of distribution) and observed increase in TCO2, assuming 50% HCO3- space of distribution as:
  Acid retention (mmoles) = [(retained HCO3-/0.5 x body wt) - observed increase in plasma HCO3-] x 0.5 bw
  Greater body acid retention is associated with faster eGFR decline. The investigators hypothesize that dietary acid reduction will lead to less acid retention.
  Comparisons among the three groups will be as follows:
  * Level at five years
  * Net change at five years

CONTACTS AND LOCATIONS:
Overall Officials: Donald Wesson, Principal Investigator — Donald E Wesson Consulting LLC

IPD SHARING:
Plan to Share IPD: Yes
Upon request, will provide study data and analysis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 90 days and for 30 days
Access Criteria: Other medical science investigators